CLINICAL TRIAL: NCT02357719
Title: Effectiveness of VistaO2 Device in Screening of Sleep Apnea/Hypopnea Syndrome
Brief Title: Effectiveness of VistaO2 FLUX Device in Screening of Sleep Apnea/Hypopnea Syndrome
Acronym: VISTAO2_FLUX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of inclusion
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Novacor (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1308191; 2014-A01733-44 (Other: AFSSAPS)
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Sleep Apnea Syndromes
Keywords: Sleep Apnea Syndromes; Polysomnography; Holter ECG; Thoracic impedance; Heart rate variability; Nasal flow
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VistaO2 FLUX device (Experimental): This device combines the transcutaneous oxyhemoglobin saturation (allowing to compute the oxyhemoglobin desaturation index), the slow variations in heart rate, the nasal flow and an index of nocturnal respiratory events calculated by analyzing the movements of the chest performed by chest impedance variations.
  Interventions: Device: VistaO2 FLUX device

INTERVENTIONS:
Device: VistaO2 FLUX device — Full night VistaO2 FLUX device monitoring synchronized with the gold standard polysomnography.
  Other Names: VistaO2 FLUX : ECG Holter recorder (Novacor, Rueil-Malmaison, France).

SUMMARY:
The high prevalence (9% in men and 4% in women) of sleep apnea / hypopnea syndrome (SAHS) in adults is now well documented as well as its cardiovascular repercussions. Previous studies showed a conclusive link between SAHS and severe cardiovascular diseases such as hypertension, myocardial infarction, heart failure and stroke.Then, SAHS is a public health issue in adults.

In this context, early detection of such a disease is crucial if the management is tailored to the patient, the practitioner's choice of therapy moving towards continuous positive airway pressure (CPAP) or mandibular advancement device. The detection is based on full nocturnal polysomnography or polygraphic recordings. Polysomnography remains the gold standard but it is a time consuming and costly examination. Polygraphic recording is a test that allows simplified the diagnosis of severe patients, but may not be sufficient for mild form of SAHS. Thus, the SAHS is a pathology under-diagnosed and under-treated. The validation of a technique for identifying patients most at risk to either limit the number of polysomnographic examination is requested.

DETAILED DESCRIPTION:
In this perspective, the development of a product screening sleep related breathing disorders for physicians, cardiologists, internists (not specialized sleep experts) would fill this need. It allows for a reliable first screening for their patients in parallel with a routine cardiological examination. Imposing a minimal human and material, the ECG Holter recorder "VistaO2 FLUX" (NOVACOR, Rueil-Malmaison, France) is a device designed to meet these requirements. This device fits into the daily management of patients with cardiac arrhythmias or sinus/atrioventricular conduction disorders, and of patients suffering myocardial infarction (arrhythmic risk stratification, detection of silent myocardial ischemia).

Analysis of heart rate variability (HRV) has already shown interest in screening SAHS. We therefore wish to evaluate the performance of the analysis of data from the screening tool VistaO2 FLUX face what the gold standard synchronized polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* sleep apnea hypopnea syndrome suspicion
* written consent

Exclusion Criteria:

* pacemaker
* diabetes
* atrial fibrillation
* electrode allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Sleep apnea hypopnea syndrome | Day 1
  Apnea hypopnea index higher than 15, evaluated by polysomnography.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ROCHE, MD-PhD, Principal Investigator — CHU de Saint-Etienne
Locations (2):
- France (2):
  - Hopital Pitié Salpetrière - APHP, Paris
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No